CLINICAL TRIAL: NCT05280067
Title: FEASIBILITY STUDY OF ZETAMET™ BONE GRAFT IN THE REPAIR OF BONE DEFECTS FROM METASTATIC BREAST CANCER IN THE SPINAL VERTEBRAL BODY: A PHASE 2A, MULTICENTER, OPEN-LABELED, SINGLE-ARM STUDY
Brief Title: ZETAMET™ BONE GRAFT IN THE REPAIR OF BONE DEFECTS FROM METASTATIC BREAST CANCER IN VERTEBRAL BONES
Acronym: ZGMBC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zetagen Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZG-2021-002
Record Dates: First submitted 2022-01-28; First posted 2022-03-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer in the Spine
Keywords: Metastatic Breast Cancer; Bone Metastases; Spine Metastases; Vancouver; Metastatic Breast Cancer to Bone; X-radiation therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Device ZetaMet™ (Experimental): ZetaMet™ is percutaneously implanted into the bone defect created by the metastatic tumor in a spinal vertebral body. ZetaMet™ is only for implantation into the vertebral body.
  Interventions: Combination Product: ZetaMet™ (ZetaFuse™ Bone Graft)

INTERVENTIONS:
Combination Product: ZetaMet™ (ZetaFuse™ Bone Graft) — ZetaMet™ (ZetaFuse™ Bone Graft) will be percutaneously implanted into the vertebral body defect(s) created by the lytic metastatic tumor.

SUMMARY:
ZetaMet™ is indicated for patients with destructive, lytic lesions due to metastatic breast cancer to bone, with or without involvement of other sites, with at least one metastatic lesion located in a vertebral body of the spine, and a Spinal Instability Neoplastic Score (SINS) ≥3 and ≤9. ZetaMet™ is percutaneously implanted into the bone defect created by the metastatic tumor in a spinal vertebral body. ZetaMet™ is only for implantation into the vertebral body.

DETAILED DESCRIPTION:
This is an open-label single-arm study. Subjects (N=10) will be recruited from up to 4 Investigational Sites in Canada. Key inclusion criteria are metastatic breast cancer to bone with at least one lytic metastatic lesion located in a vertebral body of the spine and a SINS ≥3 and ≤9. ZetaMet™ will be percutaneously implanted into the vertebral body defect(s) created by the lytic metastatic tumor. Post-operative care will be per standard of care (SOC) at the Investigational Site. Subjects will be followed for 180 days post-treatment. If post-surgical radiation treatment is planned, it should not occur for at least 84 days post-surgery to allow for bone formation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 22 (inclusive) and 75 years (inclusive) at the time of enrollment.
* Life expectancy of 12 months or more.
* Female patient with histologically confirmed diagnosis of primary breast cancer.
* Metastatic breast cancer to bone, with or without involvement of other sites (patients with single metastasis qualify)
* At least one lytic metastatic lesion located in the vertebral body of the spine.
* Normal spinal alignment.
* SINS ≥3 and ≤9.
* Signed and dated Informed Consent Form (ICF).
* Patient is willing and able to participate in required follow-up visits at the Investigational Site and to complete study procedures and questionnaires.

Exclusion Criteria:

* Vertebral body collapse.
* Spinal cord compression.
* Known allergy to Investigational Device materials.
* Using medications or any drug known to potentially interfere with bone/soft tissue healing (e.g., chronic systemic steroids).
* Current tobacco smoker or stopped smoking in past 6 months.
* Uncontrolled diabetes mellitus, HbAIC cutoff.
* An active systemic infection (e.g., hepatitis, acquired immunodeficiency syndrome (AIDS), AIDS-related complex (ARC).
* Currently participating in any investigational trial not related to this trial.
* Any other severe acute or chronic medical condition that may interfere with the interpretation of the trial results, in the judgment of the PI, which would make the patient inappropriate for entry into this trial.
* Pregnant or planning to become pregnant during the trial.

Ages: 22 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Number of Skeletal Related Events (SREs) | Day 0 up to Day 180
  SREs include pathologic fracture, spinal cord compression, radiation therapy to bone, or surgical intervention.
Number of subjects with at least one adverse event (AE) | Day 0 up to Day 180
  An AE is any unfavorable sign, symptom, or disease temporally associated with study participation, including the use of the Investigational Device and all study procedures. An AE may or may not be related to the use of the Investigational Device or a study procedure. AEs may include abnormal laboratory findings, radiologic events, medical complications, and changes from baseline in the subject's condition.
Number of subjects with at least one procedure-related AE | Day 0 up to Day 180
  A procedure-related AE is any unfavorable sign, symptom, or disease temporally associated with any study procedure. These AEs may include abnormal laboratory findings, radiologic events, medical complications, and changes from baseline in the subject's condition, related to any study procedure.
Number of subjects with at least one device-related AE | Day 0 up to Day 180
  A device-related AE is any unfavorable sign, symptom, or disease temporally associated with the Investigational Device. These AEs may include abnormal laboratory findings, radiologic events, medical complications, and changes from baseline in the subject's condition, related to the Investigational Device.
Change in SINS assessment at 21 days compared to baseline | Day 0 to Day 21 postoperatively
  The SINS is a scoring system based on six parameters; one for pain and five radiographic parameters (location, bone lesion quality, spinal alignment, vertebral body collapse and involvement of posterolateral elements). The SINS ranges 0-18. Score in range 0-6 denote stability; 7-12 intermediate instability and 13-18 instability.
Change in SINS assessment at 42 days compared to baseline | Day 0 to Day 42 postoperatively
  The SINS is a scoring system based on six parameters; one for pain and five radiographic parameters (location, bone lesion quality, spinal alignment, vertebral body collapse and involvement of posterolateral elements). The SINS ranges 0-18. Score in range 0-6 denote stability; 7-12 intermediate instability and 13-18 instability.
Change in SINS assessment at 84 days compared to baseline | Day 0 to Day 84 postoperatively
  The SINS is a scoring system based on six parameters; one for pain and five radiographic parameters (location, bone lesion quality, spinal alignment, vertebral body collapse and involvement of posterolateral elements). The SINS ranges 0-18. Score in range 0-6 denote stability; 7-12 intermediate instability and 13-18 instability.
Change in SINS assessment at 180 days compared to baseline | Day 0 to Day 180 postoperatively
  The SINS is a scoring system based on six parameters; one for pain and five radiographic parameters (location, bone lesion quality, spinal alignment, vertebral body collapse and involvement of posterolateral elements). The SINS ranges 0-18. Score in range 0-6 denote stability; 7-12 intermediate instability and 13-18 instability.
Change in Short Form 12v2 (SF-12v2) score compared to baseline | Day 0 to Day 180 postoperatively
  The 12-Item Short Form Survey version 2 (SF-12v2) is a shortened version of the SF-36v2 designed to reduce respondent burden while achieving minimum standards of precision for purposes of group comparisons involving multiple health dimensions. The SF-12v2 is given at baseline and at 180 days postoperatively.
Change in Back-specific Numeric Rating Scale for Pain (Back NRS) at 21 days compared to baseline | Day 0 to Day 21 postoperatively
  The Numeric Rating Scale (NRS) is a psychometric response scale which is commonly used in questionnaires and studies to measure the intensity of pain. In this study we will use a 11-point (0-10) scale where "0" denotes no pain and "10" is the worst imaginable pain.
Change in Back-specific Numeric Rating Scale for Pain (Back NRS) at 42 days compared to baseline | Day 0 to Day 42 postoperatively
  The Numeric Rating Scale (NRS) is a psychometric response scale which is commonly used in questionnaires and studies to measure the intensity of pain. In this study we will use a 11-point (0-10) scale where "0" denotes no pain and "10" is the worst imaginable pain.
Change in Back-specific Numeric Rating Scale for Pain (Back NRS) at 84 days compared to baseline | Day 0 to Day 84 postoperatively
  The Numeric Rating Scale (NRS) is a psychometric response scale which is commonly used in questionnaires and studies to measure the intensity of pain. In this study we will use a 11-point (0-10) scale where "0" denotes no pain and "10" is the worst imaginable pain.
Change in Back-specific Numeric Rating Scale for Pain (Back NRS) at 180 days compared to baseline | Day 0 to Day 180 postoperatively
  The Numeric Rating Scale (NRS) is a psychometric response scale which is commonly used in questionnaires and studies to measure the intensity of pain. In this study we will use a 11-point (0-10) scale where "0" denotes no pain and "10" is the worst imaginable pain.
Change in vertebral body defect size measured by CT at 42 days compared to baseline | Day 0 to Day 42 postoperatively
  Vertebral body defect size measured by CT
Change in vertebral body defect size measured by planar radiographs at 42 days compared to baseline | Day 0 to Day 42 postoperatively
  Vertebral body defect size and planar radiographs
Change in vertebral body defect size measured by CT at 180 days compared to baseline | Day 0 to Day 180 postoperatively
  Vertebral body defect size measured by CT
Change in vertebral body defect size measured by planar radiographs at 180 days compared to baseline | Day 0 to Day 180 postoperatively
  Vertebral body defect size measured by planar radiographs
Duration of use of postoperative prescription opioid | Day 180 postoperatively
  The average per group duration of intake of opioids in the post-operative setting.
Daily dose of postoperative prescription opioid use | Day 180 postoperatively
  The average per group dosage of opioids in the post-operative setting.
Naloxone concentrations in blood collected from patients at 30 minutes following the vertebroplasty procedure | 30 minutes following the placement of the surgical bandage
  Two blood samples (5 mL each) of whole blood are collected at 30 minutes following the placement of the surgical bandage (n=2 blood collections of a total of 10 mL per patient). When naloxone blood concentrations remain below 1.016-ng/mL, there is not a reduction in opioid analgesia
Naloxone concentrations in blood collected from patients at 60 minutes after the vertebroplasty procedure | 60 minutes following the placement of the surgical bandage
  Two blood samples (5 mL each) will be collected at 60 minutes following the placement of the surgical bandage (n=2 blood collections of a total of 10 mL per patient). When naloxone blood concentrations remain below 1.016-ng/mL, there is not a reduction in opioid analgesia

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - McGill University Health Center, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No